CLINICAL TRIAL: NCT05241821
Title: Management and Outcomes of Acute STROke Complicating Transcatheter Aortic Valve Implantation
Brief Title: Acute STROke Complicating TAVI - Management and Outcomes
Acronym: ASTRO-TAVI
Status: Completed | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Amos Levi, MD, Rabin Medical Center
Other Study IDs: 0502-21
Record Dates: First submitted 2022-02-05; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Stroke; Aortic Valve Stenosis; Periprocedural Complication
Keywords: periprocedural stroke; transcatheter aortic valve implantation; transcatheter aortic valve replacement
MeSH Terms: conditions — Stroke; Aortic Valve Stenosis | interventions — Fibrinolytic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conservative treatment: patients with periprocedural stroke after TAVI, treated conservatively
- Neuro-intervention: patients with periprocedural stroke after TAVI, treated with neuro-intervention
  Interventions: Procedure: Mechanical thrombectomy; Drug: Thrombolytic Agent

INTERVENTIONS:
Procedure: Mechanical thrombectomy — Percutaneous intervention aimed to retrieve/treat clot affecting the cerebral circulation.
  Groups: Neuro-intervention
Drug: Thrombolytic Agent — Drug aimed to dissolve thrombus affecting the cerebral circulation
  Groups: Neuro-intervention

SUMMARY:
Periprocedural complications of trans catheter aortic valve implantation, and particularly the occurrence of stroke has a marked impact on survival and quality of life. The characteristics of periprocedural stroke complicating TAVI, and particularly of interventions aimed to treat stroke complicating TAVI have not been systematically described. We therefore aimed is to explore the incidence and characteristics of acute stroke complicating TAVI and to describe the safety and efficacy of emergent interventions to treat acute stroke complicating TAVI.

ELIGIBILITY:
Inclusion Criteria:

* patients who have had a stroke within 30 days of TAVI

Exclusion Criteria:

* none

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with periprocedural stroke complicating TAVI
Sampling Method: Non-Probability Sample
Enrollment: 484 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-02-05 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 1-year
  All cause death
Neurologic disability free survival | 90 days
  modified rankin score (mRS) 0/1

SECONDARY OUTCOMES:
Bleeding complications | 30 days
  Severe bleeding / life-threatening bleeding as defined by VARC2 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Ran Kornowski, MD, Principal Investigator — Head of cardiology
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel